CLINICAL TRIAL: NCT07209163
Title: An Open-label, Single-arm Study Evaluating the Safety and Efficacy of Tazemetostat in Combination With Linperlisib/Golidocitinib in Patients With Relapsed/Refractory Peripheral T-cell Lymphoma
Brief Title: Combination Therapy With Tazemetostat in Relapsed and Refractory Peripheral T-cell Lymphoma
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, First Deputy Director, Hematology Department, Ruijin Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PTCL-EZH2
Record Dates: First submitted 2025-09-30; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Peripheral T Cell Lymphoma
Keywords: Peripheral T-Cell Lymphoma; Tazemetostat; Linperlisib; Golidocitinib
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — tazemetostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tazemetostat With Linperlisib (Experimental)
  Interventions: Drug: Tazemetostat; Drug: Linperlisib
- Tazemetostat With Golidocitinib (Experimental)
  Interventions: Drug: Tazemetostat; Drug: Golidocitinib

INTERVENTIONS:
Drug: Tazemetostat — Tazemetostat 800mg, twice once daily (BID), orally
Drug: Linperlisib — In Phase I, BOIN design will be adopted to enroll 3 to 12 participants, exploring the recommended Phase II dose (RP2D) at two dose levels of Linperlisib: 60 mg once daily (QD) and 60 mg QD, orally.
  In Phase II, BOP2 design will be adopted to enroll around 24 participants, aiming to evaluate the efficacy and safety of Tazemetostat with Linperlisib RP2D in patients with peripheral T-cell lymphoma with co-RHOA/TET2mut.
  Arms: Tazemetostat With Linperlisib
Drug: Golidocitinib — In Phase I, BOIN design will be adopted to enroll 3 to 12 participants, exploring the recommended Phase II dose (RP2D) at two dose levels of Lgolidocitinib: 150 mg every other day (QOD) and 150 mg QD, orally.
  In Phase II, BOP2 design will be adopted to enroll around 24 participants, aiming to evaluate the efficacy and safety of Tazemetostat with Golidocitinib RP2D in patients with peripheral T-cell lymphoma without co-RHOA/TET2mut.
  Arms: Tazemetostat With Golidocitinib

SUMMARY:
In decades, the outcome of patients with peripherial T-cell lymphomas is dismal, especially in relapsed or refractory population. After failure to the frontline treatment, patients have limited treatment options and elderly population usually have no chance to undergo transplantation due to age or comorbidity, etc. EZH2 inhibitor like Tazemetostat or SHR 2554 has been demonstrated its anti-tumor activity in PTCL either alone or in combination with other targeted agents.

This study aims to explore the efficacy and safety of Tazemetostat in combination with Linperlisib/Golidocitinib in Patients With Relapsed/Refractory Peripheral T-cell Lymphoma in the patients with peripheral T-cell lymphoma according to next-generation sequesing results.

ELIGIBILITY:
Inclusion Criteria:

1. fully understood and voluntarily signed the ICF for this study
2. aged ≥ 18 years;
3. patients with R/R PTCL who have received at least one prior systemic therapy.
4. Patients must have at least one measurable lesion by computed tomography (CT)/magnetic resonance imaging (MRI) (longest diameter of lymph node lesions > 1.5 cm or longest diameter of extranodal lesions > 1 cm); evaluable lesions: PET-CT examination showed increased local uptake in lymph nodes or extranodal sites (higher than liver) and imaging characteristics consistent with lymphoma performance
5. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 2;
6. Adequate bone marrow function, renal function, liver function: ANC ≥ 1.0 × 109/L, hemoglobin ≥ 8.0 g/dL, platelets ≥ 75 × 109/L Note: if the investigator believes that the patient 's above test values are below the lower limit of the protocol due to lymphoma invading the bone marrow, the patient can be enrolled after assessment.Creatinine clearance > 40 mL/min, calculated by Cockcroft-Gault method: • serum total bilirubin ≤ 1.5 x upper limit of normal (ULN), except for unconjugated bilirubinemia in Gilbert 's syndrome; • ALP (in the absence of bone disease), ALT, and AST ≤ 3.0 × ULN (in the presence of liver metastases, ≤ 5 × ULN); • international normalized ratio (INR) ≤ 1.5 × ULN, or activated partial thromboplastin time (APTT) ≤ 1.5 × ULN;
7. Current negative for human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV), or cytomegalovirus (CMV), and inactive if positive:

   * HBV infected patients with positive hepatitis B surface antigen (HbsAg) or hepatitis B core antibody (HbcAb)] but negative results of HBV DNA polymerase chain reaction (PCR) test can be enrolled; these patients require continuous antiviral therapy after enrollment and HBV DNA PCR test is performed every cycle;
   * Patients with positive HCV serology but negative HCV RNA test may be enrolled;
   * CMV IgM antibody positive,However, patients who tested negative for CMV DNA could be enrolled;
8. female patients of childbearing potential had to agree to use a double contraception method at least 28 days before starting study drug, during treatment, and for 6 months after the last dose of study drug, and male patients with partners of childbearing potential had to also use an effective double contraception method during the study and for 3 months after the last dose of study drug, e.g., condom, sponge plug, foam, contraceptive jelly, diaphragm cap or intrauterine contraceptive device, contraceptive pills (oral or parenteral), contraceptive implant (Implanon ®), injectable intravascular injection, or other contraceptive measures.Postmenopausal women (> 45 years of age and amenorrheic for > 1 year) and surgically sterile women are exempt from this criterion.

Exclusion Criteria:

Patients who meet any of the following exclusion criteria must be excluded from this study:

1. previously used drugs in the treatment regimen may affect the efficacy evaluation of this study (assessed by the investigator)
2. previous bone marrow malignancies, including MDS, AML, MPN, etc.
3. and have clinically significant abnormal test results as judged by the investigator;
4. inability to be orally administered, previous surgical history or severe gastrointestinal diseases such as dysphagia, active gastric ulcer, etc., which the investigator believes may affect the absorption of the study drug;
5. major surgery within 4 weeks before the first study drug administration (referring to grade 3 and 4 surgery as specified in the Measures for the Administration of Clinical Application of Medical Technology implemented on May 1, 2009);
6. current clinically significant active cardiovascular disease, such as uncontrolled arrhythmia, congestive heart failure, any grade 3 or 4 heart disease defined by the New York Heart Association functional classification, or a history of myocardial infarction within 6 months after screening.Left ventricular ejection fraction < 50% measured by echocardiography
7. Venous thrombosis or pulmonary embolism within 3 months before study drug administration;
8. History of stroke or intracranial hemorrhage within 6 months before the first study drug administration;
9. Active infection requiring systemic treatment;
10. History of inflammatory bowel disease (eg, Crohn 's disease or ulcerative colitis);
11. Known hypersensitivity to study drug;
12. Any other disease, metabolic abnormality, physical examination abnormality, or laboratory abnormality of significant clinical significance that, in the judgment of the investigator, gives reason to suspect that the patient has a disease or condition that would make the use of the study drug inappropriate or would compromise the interpretation of the study results or put the patient at high risk.
13. pregnant (positive pregnancy test) or lactating women;
14. patients who have had previous organ transplantation;
15. diagnosed or treated for malignancies other than PTCL, with the following exceptions: a) malignancies treated with curative therapy ≥ 3 years before randomization and without known active disease; b) adequately treated non-melanoma skin cancer or malignancies without evidence of disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | Tumor evaluation was assessed at screening and at the end of treatment (around 3 cycles) then every 12-24 weeks until disease progression (each cycle is 28 days) through study completion, an average of 1 year.
  Percentage of participants with complete response or partial response was determined on the basis of investigator assessments according to 2014 Lugano criteria

SECONDARY OUTCOMES:
Progression-free survival | Baseline up to data cut-off(up to approximately 2 years).
  Progression-free survival was defined as the time from the date of enrollment until the date of the first documented day of disease progression or relapse, using 2014 Lugano criteria, or death from any cause, whichever occurred first.
Complete Response Rate | Tumor evaluation was assessed at screening and at the end of treatment (around 3 cycles) then every 12-24 weeks until disease progression (each cycle is 21 days) through study completion, an average of 1 year.
  Percentage of participants with complete response was determined on the basis of investigator assessments according to 2014 Lugano criteria.
Duration of Response | Baseline up to data cut-off(up to approximately 2 years).
  Applicable to complete or partial response participants. DoR was defined as the time from the first documented date of complete or partial response until the date of the disease progression or death from any causes.
Overall survival | Baseline up to data cut-off(up to approximately 3 years).
  Overall survival was defined as the time from the date of enrollment to the date of death from any cause.
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | From enrollment to study completion, a maximum of 2 years]
  An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.